CLINICAL TRIAL: NCT00520728
Title: Efficacy of an Occupational Time Use Intervention
Brief Title: Efficacy of an Occupational Time Use Intervention for People With Serious Mental Illness
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Megan Edgelow, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OTUI1
Record Dates: First submitted 2007-08-22; First posted 2007-08-24 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Serious Mental Illness
Keywords: Schizophrenia; Psychosis; Occupational Disengagement; Occupational Imbalance
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Experimental arm receives 12 week intervention along with standard care.
  Interventions: Behavioral: Occupational Time Use Intervention

INTERVENTIONS:
Behavioral: Occupational Time Use Intervention — 12 week behavioral intervention administered by Occupational Therapists.

SUMMARY:
The purpose of this study is to test the efficacy of a new Occupational Time Use Intervention designed to increase activity participation and improve meaning in the lives of people with serious mental illness living in the community.

DETAILED DESCRIPTION:
5 Assertive Community Treatment (ACT) Teams from Kingston (n=2), Belleville (n=1), and Ottawa (n=2) will be involved in a 12 week randomized controlled trial of our Time Use Intervention. 20 subjects (4 subjects from each team) will participate in this pilot study and will be treated individually by their ACT team Occupational Therapist (1 OT per ACT Team). This pilot test will help to determine the clinical utility and efficacy of our treatment protocol.

Comparison: Standard ACT treatment with the Occupational Time Use Intervention vs. Standard ACT treatment

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-65 years of age);
* Primary diagnosis of a severe psychiatric disorder with a psychotic feature;
* Team and self-perceived occupational disengagement (low activity levels);
* Fluent in English;
* Living in a community setting and receiving ACT treatment;
* Own legal guardian (thus competent to give consent to participate), and are willing to give written informed consent to participate in the study.

Exclusion Criteria:

* Unstable mental health;
* Lack of interest in a time use intervention;
* Satisfied with current time use and occupations;
* ACT Team Occupational Therapist is subject's main Case Manager.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-08; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Change in Activity Level using a 2 day (48 hour) time use diary | Participants were tested at baseline and after 12 weeks of treatment.
Occupational Engagement using 1. 48 hour time use diary for occupational balance, 2. Engagement in Meaningful Activities Survey (EMAS) for meaning of activities, and 3. Profiles of Engagement in People with Schizophrenia (POES) to rate engagement. | Participants were tested at baseline and after 12 weeks of treatment.

SECONDARY OUTCOMES:
Clinical Utility using feedback from Therapists and Treatment Subjects | Participants were tested after 12 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Megan M Edgelow, MSc, Principal Investigator — Queen's University; Terry Krupa, PhD, Study Director — Queen's University